CLINICAL TRIAL: NCT00081952
Title: Amino Acid Therapy for Hot Flashes/Postmenopausal Women
Brief Title: Amino Acid Therapy for Hot Flashes in Postmenopausal Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: K23AT001709-01 (NIH)
Record Dates: First submitted 2004-04-27; First posted 2004-04-28 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Hot Flashes
Keywords: Postmenopause
MeSH Terms: conditions — Hot Flashes | interventions — Norleucine

INTERVENTIONS:
Drug: L-norleucine

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and effectiveness of the amino acid L-isoleucine in the treatment of hot flashes in postmenopausal women.

DETAILED DESCRIPTION:
Hot flashes affect approximately 75% of postmenopausal women. Although hormone replacement therapy (HRT) is highly effective in reducing hot flashes, long-term HRT is associated with increased rates of breast cancer and heart disease. Safe, effective, and well-tolerated hot flash therapies are needed. The amino acids L-methionine and L-isoleucine have produced reductions in hot flash frequency. However, long-term L-methionine therapy may increase cardiovascular risks. This study will evaluate the short-term effects of L-isoleucine therapy. Data from this study will be used to conduct long-term studies in the future.

Participants in this study will be randomly assigned to receive one of two different L-isoleucine doses for 2 weeks. Clinic visits will be made at baseline, Week 1, and Week 10. Participants will record the frequency and severity of their hot flashes in a diary.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Experience over 5 hot flashes per day

Exclusion Criteria:

* Hormone Replacement Therapy (HRT) in the past 2 months

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2003-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Guttuso, MD, Principal Investigator — Women's Health Initiative
Locations (1):
- Women's Health Initiative, Buffalo, New York, United States

REFERENCES:
- [Derived] Guttuso T, McDermott MP, Su H, Kieburtz K. Effects of L-isoleucine and L-valine on hot flushes and serum homocysteine: a randomized controlled trial. Obstet Gynecol. 2008 Jul;112(1):109-15. doi: 10.1097/AOG.0b013e31817d53b6. PMID 18591315